CLINICAL TRIAL: NCT01260246
Title: Sitagliptin for the Treatment of Non-alcoholic Steatohepatitis in Patients With Type 2 Diabetes.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Tisha Joy, Assistant Professor, Division of Endocrinology, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-10-533; 17389 (Registry Identifier: Office of Research Ethics, UWO)
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sitagliptin (Experimental): sitagliptin 100mg/daily for 6 months
  Interventions: Drug: sitagliptin
- placebo (Placebo Comparator): placebo match for 6 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sitagliptin — pill, 100mg/daily for 6 months
  Arms: sitagliptin
Drug: placebo — placebo match for 6 months
  Arms: placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial evaluating the impact of sitagliptin therapy in patients with concomitant type 2 diabetes and non-alcoholic steatohepatitis (NASH) on improving liver disease based on biopsy results. The effect of sitagliptin on other measures such as hormones modifying insulin release and sensitivity (termed adipocytokines), fat distribution, and biomarkers of cardiovascular risk will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Known DM2 (receiving lifestyle management and/or metformin and/or sulfonylurea
* Stable therapy for DM2 for the past 3 months
* All other medications and doses stable for past 3 months
* HbA1c 8.9% or lower (can be done in past 30 days)
* Known NASH based on the accepted American Gastroenterological Association Criteria:

  1. Alcohol consumption (< 10g/day in women and <20g/day in men)
  2. Cause of liver disease other than NAFLD (negative investigations for: viral hepatitis, iron overload, a-1 antitrypsin, ceruloplasmin, autoimmune disease)
  3. Liver histology demonstrating macrovesicular fatty change of hepatocytes, with evidence of steatohepatitis, manifested by the presence of Mallory Bodies, ballooning degeneration, lobular neutrophilic inflammation and perisinusoidal fibrosis. (If liver biopsy done within 2 years prior to screening for this trial, that biopsy will be reviewed to ensure it meets criteria for diagnosis).

Exclusion Criteria:

* Any contraindication for undergoing MRI
* Child class B or C cirrhosis
* Participation in another clinical trial
* Use of thiazoledinedione (rosiglitazone or pioglitazone) in past 6 months
* Current use of plavix
* Previous exposure to sitagliptin
* Prior history of pancreatitis
* History of anaphylaxis to another Canadian-marketed DPP-IV inhibitor (saxagliptin)
* Creatine clearance <30 ml/min
* Anaemia (haemoglobin < 110 mg/dL)
* Platelet count < 50 000 cells/mm3
* Known heart or kidney failure
* Comorbid condition that decreases natural life span (e.g. known cancer)
* Pregnant or breastfeeding or wishing to become pregnant in the next 6 months
* Current or past treatment with medications that can induce steatohepatitis (e.g. glucocorticoids, methotrexate, amiodarone etc.)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To demonstrate improvement in liver disease (based on liver biopsy)with sitagliptin. | 3 years

SECONDARY OUTCOMES:
In individuals with NASH and DM2: To document the impact of sitagliptin therapy on adipocytokines, inflammatory markers, non-traditional cardiovascular risk factors, adipose distribution, and dyslipidemia. | 3 years
In individuals with NASH and DM2: To delineate the effect of sitagliptin therapy on platelet aggregation and oxidative stress. | 3 years
In individuals with NASH and DM2: To determine the correlation between changes in histology with changes in hepatic fat demonstrated by MRI and changes in fibrosis by Fibroscan. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tisha Joy, MD, Principal Investigator — St. Joseph's Health Care, UWO
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada